CLINICAL TRIAL: NCT03655990
Title: A Prospective, Single-Centre, Post-Market Study to Evaluate the Use of Polyetheretherketone (PEEK) Full-Arch Implant-Supported Prostheses in the Edentulous Jaw
Brief Title: A Full-Arch Implant- Supported Prosthesis in the Upper and/or Lower Jaw-USA
Status: Terminated | Type: Observational
Why Stopped: Impact of COVID-19 on Recruitment
Sponsor: Juvora Ltd. (Industry)
Collaborators: PCG Clinical Services (Unknown)
Responsible Party: Sponsor
Other Study IDs: JUV17-08
Record Dates: First submitted 2018-08-08; First posted 2018-09-04 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-03

CONDITIONS: Missing Teeth
Keywords: Dentures Implant
MeSH Terms: conditions — Anodontia | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment with the JUVORA™ Dental Disc: Subjects receive the device as per normal standard practice, there are no other treatment arms for this prospective study.
  Interventions: Device: Treatment with the JUVORA™ Dental Disc

INTERVENTIONS:
Device: Treatment with the JUVORA™ Dental Disc — treatment with the JUVORA™ Dental Disc

SUMMARY:
This study follows subjects who have agreed with their dentist that their failing teeth or missing teeth all need replacing. This study follows their standard routine care with some additional assessments. The dental treatment option that replaces a whole arch or both arches (upper and lower jaws) of the mouth is call "Teeth in a Day" and information on the use of the JUVORA™ Dental Disc during this treatment is what is being collected as part of this study along with subjects follow-up care.

DETAILED DESCRIPTION:
Over the last decade full-arch metal implant-supported prosthetics have been used as a replacement for missing teeth in edentulous (toothless) patients. The standard has been a titanium metal base. Due to its potential shock-absorbing properties and patients' demands for metal-free restorations, there is rising enthusiasm surrounding the use of High Performance Polymers (HPPs) such as the polyaryletherketone (PAEKs) as metal alternatives for such cases. The JUVORA™ Dental Disc is made from PEEK-OPTIMA™ polymer (Invibio Biomaterial Solutions) which allows efficient fabrication of reliable non-metal dentures by using CAD/CAM technology to manufacture precise, custom-fit prostheses. The JUVORA™ Dental Disc is indicated for the manufacture of: full-arch implant-supported dentures and implant bars; full and partial removable dentures and overdentures; crowns and 3-unit bridges.

This study aims to evaluate the short- and long-term clinical performance and patient satisfaction of the JUVORA™ full-arch implant-supported prostheses.

Two subjects will be included in a run-in phase and 10 subjects will be included in the main study.

The subjects will be followed-up at 6 weeks, 6 months, 12 months and for as long as willing yearly after the implant of the definitive prosthesis (artificial teeth).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older in need of a full-arch implant supported rehabilitation in a single jaw (mandibular or maxillary) or both edentulous jaws (mandibular and maxillary).
* Subjects with adequate bone quality and quantity to allow the placement of a minimum of four Neodent implants into the arch area.
* Subjects who, in the opinion of the Investigator, are able to understand this clinical study, co-operate with the procedures and are willing to return to the clinic for all the required post-operative follow-ups.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical study and from whom consent has been obtained.

Exclusion Criteria:

Female subjects who are pregnant or lactating.

* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects with any condition that would compromise their participation and follow-up in this clinical study.
* Subjects with insufficient bone volume or quality in the edentulous jaw.
* Subjects on any chemotherapeutic or bisphosphonate medications.
* Subjects with evidence of tumour and/or malignant disease with resultant life expectancy of less than 2 years.
* Subjects who smoke more than 10 cigarettes per day.
* Subjects who are currently enrolled in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated to receive a full-arch implant-supported prosthesis in a single jaw (mandibular or maxillary) or full-arch implant-supported prosthesis in both jaws (mandibular and maxillary).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Survival of the Prosthetic | 12 months
  Survival will be evaluated using the ITI Treatment Guide Volume 8 - Survival is defined as "is the prosthesis present in the mouth at the time of assessment ("presence or absence")

SECONDARY OUTCOMES:
Patient quality of life assessment using a patient questionnaire. | 6 weeks 6 & 12 months
  Overall health-related QOL questionnaires - (Oral Health Impact Profile) OHIP - 14 measures peoples perceptions of the social impact of Oral Disorders on their well-being. Fourteen questions with 5 possible answers: Never, Hardly Ever,Occasionally, Fairly Often, Very Often. Questions are related to whether subjects have had problems with their teeth, mouth or dentures.
Oral and dental:Patients will be assessed for a history of Bruxism (grinding of the teeth). | 6 weeks 6 &12 months
  If patients have suffered with Bruxism they will be asked if they have been wearing their night guard during their dental treatment.
Oral and dental: Patients will be checked for occlusion. | 6 weeks &12 months
  This is a way of checking when the teeth are clenched how many generalized number of contacts there are between the two arches (i.e., how many teeth are in contact between the upper and lower jaw arches)
  * Amount of cantilever from the most distal implant for the left side will be recorded in (mm)
  * Amount of cantilever from the most distal implant for the right side will be recorded in (mm)
Survival of the implant in the patients mouth. | 12 months
  Survival will be evaluated in accordance with the ITI Treatment Guide Volume 8. Survival is defined as 'is the implant present in the mouth at the time of the assessment' (presence or absence).
Success of the implant in the patients mouth. | 12 months
  Success will be evaluated in accordance with the ITI Treatment Guide Volume 8. Implants will be deemed to be successful if they are present:without implant fracture, without radiolucency changes from pre-treatment condition, without mobility, without pain, infection (suppuration, abscess and/or fistula), or paresthesia and without bone loss > 2mm.
Success of the implant in the patients mouth according to marginal bone resorption. | 12 months
  Success will be evaluated according to the marginal bone resorption (bone loss). Evaluated using a conventional digital panorex xray and measured. The measurements will be performed on the mesial and distal aspects of the implant platform and the lowest value will be recorded.
Success of the implant in the patients mouth according to the presence of Peri-implantitis. | 12 months
  Success will be evaluated according to the presence of Peri-implantitis (presence of inflamed mucosa with positive bleeding on probing and or suppuration ≥5mm and cumulative bone loss of ≥ 2mm and/or ≥3 threads of implant)
Success of the implant in the patients mouth according to modified plaque index (mPI). | 12 months
  Success will be evaluated according to the Modified Plaque Index (mPI) will be evaluated by inserting a periodontal plastic probe 1 mm into the peri-implant sulcus running a circular movement all around the implant and measured in a scale between 0 to 3:
  0 = no detection of plaque
  1. = plaque only recognized by running a probe across the smooth marginal surface of the implant
  2. = plaque can be seen by the naked eye
  3. = abundance of soft matter
Success of the implant in the patients mouth according to Modified Bleeding Index (mBI). | 12 months
  Success will be evaluated according to the Modified Bleeding Index (mBI) evaluated by inserting a periodontal plastic probe 1 mm into the peri-implant sulcus running a circular movement all around the implant and measured in a scale between 0 to 3:
  0 = no bleeding when a periodontal probe is passed along the mucosal margin adjacent to the implant
  1. = isolated bleeding spots visible
  2. = blood forms a confluent red line on mucosal margin
  3. = heavy or profuse bleeding
Success of the implant in the patients mouth according to the probing depth. | 12 months
  Success will be evaluated according to the Probing Depth. The depth of the peri-implant sulcus will be determined by measuring the distance from the mucosal margin to the base of the sulcus using a calibrated periodontal probe using minimal force (< 0.3M).
Success of the implant in the patients mouth according to Soft Tissue Reactions. | 12 months
  Success will be evaluated according to Soft Tissue Reactions. The presence or absence of oral mucosal disorders not related to peri-implant infection (e.g., reporting of allergic reactions, lichen planus) will be recorded.
Success of the implant in the patients mouth according to Mechanical Complications. | 12 months
  Complications related to the implant include implant fracture, abutment/screw fracture and loosening will be reported.
Success of the prosthesis assessed according to specific criteria and in accordance with the ITI Treatment Guide Volume 8. | 12 months
  Success will be evaluated in accordance with the ITI Treatment Guide Volume 8. JUVORA™ prosthesis will be deemed to be successful if they are present:
  * without complications (fracture of the veneering material, framework fracture and loss of retention of the prosthesis)
  * with adequate 'in-mouth comfort': using a grading system between 0 (poor) and 10 (excellent).
  * with adequate function (chewing): Function is defined as the chewing ability of the patient to chew different food types (meat, fruit, vegetables, salad) using a grading system between 0 (poor) and 10 (excellent).
  * with adequate aesthetics: Aesthetic examination including surface luster and staining, colour stability, translucency, and anatomic form.
  Also Attachment Performance:
  Attachment performance will involve examination and recording of any issues related to attachment performance (presence or absence).
Device Deficiencies reported for the JUVORA™ Dental Disc/prosthesis only: Inadequacy of medical device with respect to identity, quality, durability, reliability, safety and performance and includes malfunctions, user errors and inadequate labelling. | 6 weeks 6 & 12 months
  Device Deficiency data collected:
  1. Date deficiency occurred, if it could have led to a medical occurrence:
     if either a suitable action had not been taken or if intervention had not been made or if circumstances had been less fortunate
  2. If could have led to a Serious Adverse Device Effect (SADE)?
  Which is a serious adverse event according to one of the criteria below and device related:
  Results in death Is life-threatening Requires inpatient hospitalisation or prolongation of existing hospitalisation Results in persistent or significant disability/incapacity (including a medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function or permanent impairment to a body structure or a body function) Is a congenital anomaly/birth defect
Patient adverse events related to the dental surgery and treatment only will be collected. | 6 weeks 6 & 12 months
  Information collected will be as follows:
  date and time of onset whether it is mild, moderate or severe. the frequency and the action taken.
  If it is related to the device and if so, is it anticipated or serious and when or if it is resolved.
If the patient has to have any additional dental procedures and or treatments will be collected. | 6 weeks 6 & 12 months
  The reason for the additional dental procedure treatments will be collected along with the date and broken down under the following reasons:
  Failed Implant Severe Bone Loss Loss of Attached Tissue

OTHER OUTCOMES:
Technical Satisfaction not related to the patient | between 4 - 6 months prior to fixture in the patients mouth.
  Data collected during the Laboratory processing of the JUVORA™ Dental Disc into the prosthesis.
  Infrastructure manufacturing issues? Framework integrity issues? Veneer adhesion issues?

CONTACTS AND LOCATIONS:
Overall Officials: Juvora, Study Director — Juvora Ltd.
Locations (1):
- Dr Robert Lemke, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study location web site for enquiries — http://oralsurgerytx.com